CLINICAL TRIAL: NCT01825928
Title: Randomized, Double-blind, Placebo-controlled Trial of Paliperidone Extended-Release Tablets for The Treatment of Methamphetamine Dependence in Chinese Patients After Detoxification
Brief Title: An Study of Paliperidone Extended-Release Tablets in the Treatment of Methamphetamine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Hao (Other)
Responsible Party: Sponsor-Investigator, Wei Hao, The Second Xiangya Hospital of Cental South University, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100000-068944
Record Dates: First submitted 2013-03-28; First posted 2013-04-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; paliperidone
MeSH Terms: interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paliperidone (Experimental): paliperidone arm,3mg/pill,3mg/day.last84 days.
  Interventions: Drug: Paliperidone
- placebo (Placebo Comparator): placebo group,3mg/pill,3mg/day non-forced titration method,last84 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Paliperidone — Paliperidone group,3mg/pill,3mg/day forced titration method,last 84 days
  Other Names: Paliperidone Extended-Release Tablets; Invega
  Arms: paliperidone
Drug: placebo — placebo group,3mg/pill,3mg/day forced titration method,last 84 days
  Arms: placebo

SUMMARY:
Methamphetamine substance use is common worldwide. No approved pharmacologic treatments for methamphetamine dependence exist. paliperidone are Second generation antipsychotics，and have effects of blocking dopamine2(D2) and 5-hydroxytryptamine 2A(5-HT) receptors neurotransmitters.To determine whether mirtazapine would reduce methamphetamine use among methamphetamine addicts.

DETAILED DESCRIPTION:
Methods:A Multiple-Center, Randomized, Double-Blind.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years to 60 years
* Met the Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria for METH dependence with psychosis
* Completing inpatient METH detoxification (≤30 days) with psychotic symptoms disappeared
* Beoff any anti-psychotic medication for 7 days after discharging from hospital were enrolled at clinical site
* Participants were interesting in reducing or stopping METH use
* Every patient also had a significant other (eg., spouse or relative) who supervised their compliance with the visit schedule and study procedures
* Women of childbearing potential agreed to use contraception during the study.

Exclusion criteria:

* Pregnancy or breastfeeding;
* Significant medical conditions (eg., acute renal failure, endocarditis, and tuberculosis); hepatic failure; past or present history of an AIDS-indicator disease; active hepatitis or aspartate amino transferase or alanine aminotransferase more than three times the upper limit of normal
* Known intolerance or hypersensitivity to paliperidone ER; other psychosis; present dependence on substances other than METH or poly-substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Abstinent time of Methamphetamine addict | up to 84 days
  The outcome was the confirmed abstinence during 12 weeks. Confirmed abstinence was defined as a negative urine drug test. The following aggregate measures of urine drug test results were calculated: the time-to-first positive urine test, the Treatment Effectiveness Score (TES; the sum of the number of METH-free urine samples submitted per participant ), the longest period of MA abstinence during the 84 days.

SECONDARY OUTCOMES:
Time (day) to first psychosis relapse from baseline to 84 days | up to 84 days
  psychosis assessement was made once a week.Psychotic symptom relapse was defined as one or more of the following: (1) hospitalization for psychotic symptoms; deliberate self-injury or violent behavior, or suicidal or homicidal ideation that was clinically significant;25% increase in PANSS total score;for patients who scored >40 at randomization, or a 10-point increase for patients who scored ≤40 at randomization for two consecutive assessments (within 1 week), and (4) increase in prespecified individual PANSS items scores (P1, P2, P3, P6, P7 and G8) to ≥5 for patients whose score was ≤3 at randomization, or to ≥6 for patients whose score was 4 at randomization for two consecutive assessments (within 1 week)
Change from baseline in CGI-S scores at 84 days | up to 84 days
  general condition assessment was made by CGI-S once a week, and calculated the total scores
Change from baseline in Visual Analogue Scale (VAS) at 84 days | up to 84 days
  Methamphetamine craving assessment was made by VAS once a week, and calculated the total scores
number of treatment day which calculated from randomization to the last visiting point | up to 84 days
  record the follow up time

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hao, MD., Ph.D., Study Director — Central South University
Locations (1):
- The Second Xiangya Hospital of Central University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided